CLINICAL TRIAL: NCT07036211
Title: Transmission of Oncogenic HPV Infection Among Families
Acronym: TREVINO
Status: Not yet recruiting | Type: Observational
Sponsor: Tampere University Hospital (Other)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: R23092
Record Dates: First submitted 2025-04-23; First posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Human Papilloma Virus (HPV); Cervical Carcinoma; Oropharyngeal Carcinoma; Transmission Vertical; Transmission; Human Papillomavirus Infection
Keywords: Oropharyngeal cancer; Cervical cancer; HPV
MeSH Terms: conditions — Uterine Cervical Neoplasms; Oropharyngeal Neoplasms; Papillomavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will take swab/brush samples from the oral cavity, and cervix/vagina/anus (women), additionally urine (men) as well as saliva samples and gargle samples from oral cavity from all participating. The follow-up samples are self-collected samples: saliva, oral gargle, genital/urine sample. From the offspring the oral gargle and saliva is collected at each follow-up visit with optional vagina and urine sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with HPV associated disease: 1) colposcopy clinic detected persisting HR-HPV infection, 2) diagnosed cervical cancer; or 3) diagnosed Oral squamous cell carcinoma (OSCC).
- Offspring of patients with HPV associated disease: Children over 12 years old
- Sexual partner (spouse) of patients with HPV associated disease: Women or men

SUMMARY:
The goal of the Transmission of Oncogenic HPV Infection Among Families (TREVINO) study is to improve understanding of how high-risk human papillomavirus (HPV) infections are transmitted within families. The research focuses on transmission between sexual partners and between parents and children. It also examines how the various microbes may influence the persistence of HPV infections and the development of HPV-related cancers.

The study will include up to 300 couples recruited from gynecology and ear, nose, and throat (ENT) clinics in Finland, as well as their children. Participants include individuals with persistent HPV infection, cervical precancer or cancer, or HPV-related head and neck cancer, along with their partners and potentially their offspring.

Participants will provide self-collected samples from the oral and genital areas at multiple time points over up to five years. Questionnaires addressing medical, behavioural, and environmental factors will be completed.

The study is conducted at Tampere University Hospital and Kuopio University Hospital in Finland. Results will inform HPV screening and prevention programs, improve understanding of family-level transmission, and identify potential microbial and genetic markers linked to cancer risk.

DETAILED DESCRIPTION:
TREVINO (Transmission of Oncogenic HPV Infection Among Families) is a prospective and longitudinal research project aimed at investigating the transmission, persistence, and clinical consequences of high-risk human papillomavirus (HPV) infections within family. The study also explores how various microbes, as well as genetic and environmental factors, influence HPV infection outcomes.

The study consists of three main parts:

Part 1 focuses on assessing the prevalence, concordance and transmission of HPV infections among individuals with HPV-associated precancerous or cancerous lesions and their sexual partners (spouses).

Part 2 aims to characterize the role of the microbes in HPV persistence and the progression to cervical and oropharyngeal cancer.

Part 3 investigates vertical and horizontal transmission of HPV and microbial communities within families by including offspring.

Participants will include up to 300 couples recruited from Tampere University Hospital and Kuopio University Hospital in Finland, as well as their children. Recruitment targets women or men attending gynecology or ENT clinics with confirmed persistent HPV infection, cervical precancer or cancer, or oropharyngeal squamous cell carcinoma (OSCC). Partners are invited to participate regardless of symptom status.

Samples will be collected from patients with HPV associated decease at baseline, and then at 6, 12, and 24 months, with extended follow-up to 60 months for individuals with persistent infections. Self-sampling kits for oral, genital, urine, saliva, and gargle samples will be distributed and returned via mail. Partners will give samples at 0, 12 and 24 months and will have the extended follow-up for individuals with persistent infections. Children will provide oral samples, and optional urine or vaginal samples at 0, 12 and 24 months. Offspring over 30 years old will also have the opportunity to participate the extended follow-up.

Biological assays include HPV genotyping, HLA typing, immunohistochemistry, in situ hybridization, metagenomic sequencing, methylation analysis, and targeted sequencing.

Statistical analysis plans will vary by study objective and will include logistic regression, generalized estimating equations (GEE), ROC curve construction, and compositional methods for microbial profiling. All analyses will be conducted using Stata.

The study has been approved by the Pirkanmaa County Ethical Review Board. Recruitment is expected to begin in spring 2025. Findings will support the development of prevention strategies, improved risk stratification, and innovative diagnostic and therapeutic approaches for HPV-associated diseases.

ELIGIBILITY:
Inclusion Criteria:

* Patient with colposcopy clinic detected persisting HR-HPV infection
* Patient with diagnosed cervical cancer
* Patient with diagnosed OSCC
* Patients' sexual partners of women or men that are referred to the colposcopy/gynecological oncology/ENT
* offspring (over 12 years old) of the referred couples

Exclusion Criteria:

* Candidate who don't speak Finnish

Ages: 12 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients who will be attending either the ObGyn or ENT at Tampere University Hospital (TAUH) or at Kuopio University Hospital (KUH) concerning HPV associated decease and their spouses and offspring.
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2027-05 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
HPV genotype among patients with HPV associated disease and their sexual couples | From enrollment to 24 month follow-up samples
  All oral and genital samples are genotypes using extended HPV genotyping assays that detect at least 25 different HPV genotypes separately.

CONTACTS AND LOCATIONS:
Overall Officials: Karolina Louvanto, Professor, Principal Investigator — Tampere University
Locations (2):
- Finland (2):
  - Kuopio University Hospital, Kuopio
  - Tampere University Hospital, Tampere

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Time Frame: Beginning 3 months after publication with no end date
Access Criteria: IPD that underlie the results reported in a publication, after de-identification, will be available for researchers who provide a methodologically sound proposal with achievable aims. Proposals should be directed via e-mail to the PI of the study (KL); data requestors will need to sign a data access agreement.